CLINICAL TRIAL: NCT00676598
Title: A Prospective Analysis of the Effect of Therapeutic Hypothermia After Cardiac Arrest
Status: Completed | Type: Observational
Sponsor: Advocate Hospital System (Other)
Responsible Party: Principal Investigator, Christine Kulstad, Attending Physician, Advocate Hospital System
Other Study IDs: AHCIRB 4305
Record Dates: First submitted 2008-05-12; First posted 2008-05-13 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Cardiac Arrest
Keywords: therapeutic hypothermia
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Therapeutic hypothermia has been shown to improve survival and neurologic outcome in patients resuscitated after ventricular fibrillation arrest.

Few studies have examined whether therapeutic hypothermia is effective outside the research setting, or with other presenting rhythms.

Our institution, a large community teaching hospital, instituted a therapeutic hypothermia protocol in November 2006 for all resuscitated cardiac arrest patients.

The investigators seek to determine the mortality rate of our protocol and compare our complication rates with those of previously published studies.

DETAILED DESCRIPTION:
The use of therapeutic hypothermia has been shown to have a beneficial effect on neurologic outcomes of patients resuscitated from cardiac arrest in a limited number of clinical sites. Based on available data, current recommendations from the American Heart Association include a level 2a endorsement of therapeutic hypothermia for cardiac arrest from ventricular fibrillation with persistent coma, and a level 2b recommendation for cardiac arrest from any other rhythm. To date there have been no formal studies presented that demonstrate an improvement in outcome when a hypothermic protocol is implemented in a community hospital. The investigators plan to prospectively collect data on patients enrolled in the therapeutic hypothermia protocol to evaluate clinical outcomes and compare these outcomes with historic controls, with the hypothesis that patients enrolled in the hypothermic protocol will have improved neurologic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Any adult non-pregnant patient who is unresponsive after resuscitation from cardiac arrest regardless of presenting rhythm and who survives to hospital admission.

Exclusion Criteria:

* hypotension (SBP <90), initial temperature < 30 °C, trauma, primary intracranial event, or active coagulopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any adult non-pregnant patient who is unresponsive after resuscitation from cardiac arrest regardless of presenting rhythm and who survives to hospital admission.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2007-01; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erik B Kulstad, MD,MS, Study Chair — advocate christ medical center
Locations (1):
- Adcovate Christ Hospital, Oak Lawn, Illinois, United States